CLINICAL TRIAL: NCT01881464
Title: Anti TNF α Improves Endothelial Dysfunction in IBD Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CMC-13-0006-CTIL
Record Dates: First submitted 2013-06-11; First posted 2013-06-19 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2013-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CRP, CBC,Serum for future metabolomics perpus.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- endothelial dysfunction assessment: This study is a one arm study . In this arm we will assess endothelial function (with Endopath device) in patients with Crohn's disease, before and after treatment of anti TNF α and other medication, and evaluate the possible role of tumor necrosis factor (TNF)-α in the pathophysiology of this abnormality.
  Interventions: Device: Endopath from Itamar medical - FDA approved device.; Drug: Anti TNF Alfa.

INTERVENTIONS:
Device: Endopath from Itamar medical - FDA approved device. — endothelial function assessment by Endopath device
Drug: Anti TNF Alfa. — This study will assessed the presence of endothelial dysfunction in patients with Crohn's disease before and after 12 weeks treatment of anti TNF α.
  Other Names: HUMIRA-ADALIMUMAB, REMICADE-INFLIXIMAB

SUMMARY:
Study hypothesis - this study will assess the presence of endothelial dysfunction in patients with Crohn's disease before and after 12 weeks treatment of anti TNF α.

DETAILED DESCRIPTION:
Crohn's Disease (CD) is a life long disease that mainly affects young adults. There is evidence That gut tissue injury is the result of an abnormal immune response that involved multiple non immune cellular systems including the intestinal microvascular endothelial cell. Moreover, clinical studies have shown that 1-7% of irritable bowel disease (IBD) patients suffer from arterial and venous thromboembolic complication.

Chronic inflammation has a major role in the development and propagation of endothelial dysfunction, which can lead to coronary artery disease.

Endothelial dysfunction has been described in patients with various and diverse chronic inflammatory conditions. Over the last few years, dysfunction of vascular endothelium has been widely recognized as the first step in the development of atherosclerosis. Several inflammatory mediators, such as C-reactive protein (CRP), Tumor Necrosis Factor α, (TNF α), nitric oxide (NO), vascular endothelial growth factor, CD-40, interleukin-6 (IL-6), which are up-regulated in IBD, also are known to impact vascular impact.

The normal endothelium produces a vasodilatatory response to ischemia referred to us as reactive hyperemia. Shear stress on the blood vessel wall leads to the production and release vasodilatation. With endothelial dysfunction there is often either a blunted vasodilatatory in response to ischemic event, and chronic inflammation.

The hypothesis of this study is that patients with Crohn's disease have an increased incidence of endothelial dysfunction, which can be corrected or improved by treatment with anti TNF α.

The purpose of our study was to assess endothelial function in patients with Crohn's Disease, before and after treatment (steroids, immunomodulators, and anti TNF α). This study assessed the presence of endothelial dysfunction in patients with Crohn's disease and evaluated the possible role of tumor necrosis factor (TNF)-α in the pathophysiology of this abnormality.

In this study we will preformed an endothelial function test before and after treatment by Endopath device from Itamar medical, FDA approved.

Safety- Each subject will be screened by clinical history, physical examination, electrocardiogram, chest X-ray, Mantoux test (PPD), routine chemical analysis, and biomarkers.

The study protocol has been approved by the local institutional review board.

ELIGIBILITY:
Inclusion Criteria:

* Non smoker
* No history of IHD or other known risk factors for IHD

Exclusion Criteria:

* Patients who had been treated with anti TNF α 4 weeks before the study
* As well as those who received corticosteroids within 1 week before the study.
* DM, IHD, CRF, SMOKER

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: IBD Patients.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
This study will assessed the presence of endothelial dysfunction in patients, C with crohn's disease before and after 12 weeks treatment of anti TNF α. CDAI, CRP. | 12 month
  In this study we will preformed an endothelial function test before and after 12 weeks of treatment, by Endopath device from Itamar medical, FDA approved.
  Endo-PAT tests can be carried out in both the office and hospital settings, with patients positioned either sitting or supine. Endo-PAT bio-sensors are placed on the index fingers of both arms. The test takes 15 minutes to complete, is very easy to perform, and is both operator and interpreter independent. Thermo-neutral, quiet surroundings are recommended. Endo-PAT quantifies the endothelium-mediated changes in vascular tone, elicited by a 5-minute occlusion of the brachial artery (using a standard blood pressure cuff).

CONTACTS AND LOCATIONS:
Overall Officials: Zittan Eran, Principal Investigator — CARMEL MEDICAL CENTER - HAIFA -ISRAEL
Locations (1):
- Carmel Medical Center, Haifa, Israel